CLINICAL TRIAL: NCT03230019
Title: Two-Lumen Catheterization Versus Chest Tube Placement in Patients With Lung Wedge Resection: A Prospective Randomized Trial
Brief Title: Two-Lumen Catheterization For Lung Wedge Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wen-zhao ZHONG (Unknown)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Wen-zhao ZHONG, Guangdong General Hospital, Guangdong Provincial People's Hospital
Organization: GuangdongPPH (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBL-1
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Thoracic Surgery, Video-Assisted
Keywords: wedge resection; tubeless
MeSH Terms: interventions — Chest Tubes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chest tube (Active Comparator): VATS with chest tube placement
  Interventions: Procedure: chest tube
- two-lumen catheter (Experimental): VATS with two-lumen catheterization
  Interventions: Procedure: two-lumen catheterization; Device: two-lumen catheter

INTERVENTIONS:
Procedure: chest tube — VATS with chest tube placement
  Arms: chest tube
Procedure: two-lumen catheterization — VATS with two-lumen catheterization long the midclavicular line, second intercostal space
  Arms: two-lumen catheter
Device: two-lumen catheter — central venous catheter(two-lumen 7-Fr-20cm)
  Arms: two-lumen catheter

SUMMARY:
This study evaluates the viability and safety of two-lumen catheterization versus chest tube placement in patients with lung wedge resection. Half of participants will receive routine chest tube placement, while the other half will receive a two-lumen central venous catheterization along the midclavicular line, second intercostal space for remedial gas-remove.

DETAILED DESCRIPTION:
With the development of video-assisted thoracoscopic surgery (VATS) techniques, minimally invasive thoracic surgery has evolved considerably over the last three decades. The concept of "tubeless" involves non-intubated anesthesia with spontaneous ventilation and no chest tube placement. Chest tube placement always causes pain, and its duration is known to be one of the most important factors influencing hospital stay and costs. Early tube removal allows patients to breathe deeply with less pain, which leads to more compliance with chest physiotherapy, as demonstrated by a concomitant improvement in patients' ventilatory function. Hence, more and more experienced surgeons choose the omission of chest tube placement after lung wedge resection. However, based on previous retrospective studies, residual pneumothorax was noted in about 10~40% cases, and some of them need re-intervention. Hence, the investigators designed a intra-operative two-lumen catheterization for remedial gas-remove. Therefore, this study evaluates the viability and safety of two-lumen catheterization versus chest tube placement in patients with lung wedge resection.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative radiology revealed solitary peripheral pulmonary nodule, with both size and depth less than 3 cm
2. Lung wedge resection for tumor biopsy to elucidate drug resistant mechanism or confirm diagnosis

Exclusion Criteria:

1. Previous ipsilateral thoracic surgery or extensive adhesion
2. Preoperative radiology revealed pneumonia or atelectasis
3. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
4. Bleeding tendency or anticoagulant use
5. Pregnancy or breast feeding
6. Patient who can not sign permit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative adverse event incidence rate | 1 months
  To evaluate the incidence rate of pneumothorax (a pneumothorax greater than 2.0 cm on X-ray) or pleural effusion (>800ml) in both groups.
Length of post-operative hospital stay | 1 week
  To evaluate the length of post-operative hospital stay
Rate of post-operative related complications | 1 week
  To evaluate the rate of post-operative related complications within 7 days of surgery

SECONDARY OUTCOMES:
Postoperative pneumoderm incidence rate | 3 days
  To evaluate the postoperative pneumoderm incidence rate in both groups.
The time of post-operative extubation | 1 week
  To evaluate the time of duration of chest tube or catheterization.
Postoperative pulmonary function recovery | 1 week
  To evaluate the postoperative cardiopulmonary function recovery via 6-minute walk test in both groups.
Postoperative pain score | 1 day
  To evaluate the pain score via NRS pain scale first day after surgery.
Postoperative wound satisfaction | 1 month
  To evaluate the post-operative wound healing condition .

OTHER OUTCOMES:
Characteristics of plasma exosome for the solitary pulmonary nodules | 1 month
  We prospectively collect the preoperative plasma sample of patients with solitary pulmonary nodule in this study to determine the diagnostic value and molecular characteristics of plasma exosome-derived miRNAs for these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Zhao Zhong, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang SM, Wang ML, Hung MH, Hsu HH, Cheng YJ, Chen JS. Tubeless Uniportal Thoracoscopic Wedge Resection for Peripheral Lung Nodules. Ann Thorac Surg. 2017 Feb;103(2):462-468. doi: 10.1016/j.athoracsur.2016.09.006. Epub 2016 Nov 16. PMID 27865474
- [Background] Watanabe A, Watanabe T, Ohsawa H, Mawatari T, Ichimiya Y, Takahashi N, Sato H, Abe T. Avoiding chest tube placement after video-assisted thoracoscopic wedge resection of the lung. Eur J Cardiothorac Surg. 2004 May;25(5):872-6. doi: 10.1016/j.ejcts.2004.01.041. PMID 15082297
- [Background] Ueda K, Hayashi M, Tanaka T, Hamano K. Omitting chest tube drainage after thoracoscopic major lung resection. Eur J Cardiothorac Surg. 2013 Aug;44(2):225-9; discussion 229. doi: 10.1093/ejcts/ezs679. Epub 2013 Jan 12. PMID 23313864
- [Derived] Wei S, Zhang G, Ma J, Nong L, Zhang J, Zhong W, Cui J. Randomized controlled trial of an alternative drainage strategy vs routine chest tube insertion for postoperative pain after thoracoscopic wedge resection. BMC Anesthesiol. 2022 Jan 18;22(1):27. doi: 10.1186/s12871-022-01569-w. PMID 35042458
- [Derived] Zhang JT, Qin H, Man Cheung FK, Su J, Zhang DD, Liu SY, Li XF, Qin J, Lin JT, Jiang BY, Song Dong, Liao RQ, Qiang N, Yang XN, Tu HY, Zhou Q, Yang JJ, Zhang XC, Zhang YN, Wu YL, Zhong WZ. Plasma extracellular vesicle microRNAs for pulmonary ground-glass nodules. J Extracell Vesicles. 2019 Sep 18;8(1):1663666. doi: 10.1080/20013078.2019.1663666. eCollection 2019. PMID 31579436